CLINICAL TRIAL: NCT04098406
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study in Early Symptomatic Amyotrophic Lateral Sclerosis Patients on Stable Background Therapy to Assess Bioenergetic Catalysis With CNM-Au8 to Slow Disease Progression in ALS.
Brief Title: Therapeutic Nanocatalysis to Slow Disease Progression of Amyotrophic Lateral Sclerosis (ALS)
Acronym: RESCUE-ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clene Nanomedicine (Industry)
Collaborators: Clene Australia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNMAu8.205
Expanded Access: NCT04081714 (Temporarily not available)
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Gold; Nanocrystal; electromyography; ALS; Nanoparticle
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, parallel group, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The drug formulations were identical in appearance (size, shape, volume, color) and smell. The packaging and labeling were designed to maintain blinding to the Investigator's team and to patients. There are no visible differences between the active drug, and placebo dosing units
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The matched placebo used in this study consisted of water, sodium bicarbonate, and food coloring to match volume and color of the experimental treatment
  Interventions: Drug: Placebo
- 30 mg CNM-Au8 (Experimental): 30mg suspension of clean-surfaced, faceted, gold nanocrystals in 60ml of sodium bicarbonate buffered water
  Interventions: Drug: CNM-Au8

INTERVENTIONS:
Drug: CNM-Au8 — CNM-Au8 is a dark red/purple-colored liquid formulation consisting of a stable suspension of faceted clean surfaced elemental gold nanocrystals in buffered deionized water with a nominal concentration of 0.5 mg/mL of gold. The formulation is buffered by sodium bicarbonate present at a concentration of 0.546 mg/mL. There are no other excipients. The drug product is formulated to be taken orally and will be provided in single dose 60 mL HDPE containers.
  Arms: 30 mg CNM-Au8
Drug: Placebo — Placebo was liquid with identical color and taste
  Arms: Placebo

SUMMARY:
The objective of this trial was to assess the efficacy, safety, and PK/PD effects of CNM-Au8 as a disease-modifying agent for the treatment of ALS by utilizing electrophysiological measures to detect preservation of motor neuron function. The primary endpoint was the mean change in the average difference between active treatment and placebo from Baseline through Week 36 evaluated by electromyography.

DETAILED DESCRIPTION:
This was a multi-centre randomized, double-blind, parallel group, placebo-controlled study of the efficacy, safety, pharmacokinetics, and pharmacodynamics of CNM-Au8 in patients who are newly symptomatic within 24-months of Screening and with a clinically probable or possible or definite ALS diagnosis per the Awaji-Shima criteria.

Patients were screened over up to a 6-week period. Patients who met the inclusion criteria and none of the exclusionary criteria were enrolled into the clinical study. Patients were randomized 1:1 into one of two groups: either active treatment with CNM-Au8 30 mg or Placebo.

All patients received their randomized oral treatment daily over thirty-six (36) consecutive weeks during the Treatment Period.

There were up to four study periods:

1. Up to a six (6) week screening period (Screening Period);
2. A thirty-six (36) week blinded randomized treatment period (Treatment Period);
3. Up to a forty-eight (48) week optional open-label extension period (Open-Label Period);
4. A four (4) week safety follow-up period following completion of either the Treatment or Open-Label period or in the case of Early Termination (Safety Follow-Up Period).

Per protocol, all patients received their blinded and randomized oral treatment daily over at least 36 consecutive weeks during the Treatment Period.

For those patients not transitioning into the optional OLE period, patients completed a safety follow-up visit 4-weeks following study drug discontinuation.

An independent DSMB was responsible for monitoring the safety of the study on a quarterly basis and ad hoc at the request of the DSMB or the Sponsor (e.g., in the event of unexpected SAEs) to review data throughout the Treatment Period. The DSMB may make recommendations on the conduct of the study, including study termination. Appropriate procedures will be detailed in a DSMB Charter.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and give written informed consent.
2. Male or female patients aged 30 years or greater (inclusive) and less than 80 years of age at the time of Screening.
3. Patients whose conditions are defined as possible or probable or definite ALS per the diagnostic criteria by Awaji-Shima criteria as determined by a neurologist sub- specialising in ALS (e.g., the Principal Investigator by study site).
4. For patients taking riluzole, stable dosing of riluzole over the prior 30-days from Screening.
5. At the time of Screening either disease duration less than or equal to 24-months from symptom onset, or disease duration less than or equal to 12-months from diagnosis.
6. Forced vital capacity (FVC) 60% of predicted value as adjusted for gender, height, and age at the Screening Visit.
7. Patient who has established care with a neurologist at one of the specialized ALS clinics involved in the study and will maintain this clinical care throughout the study. If a patient is referred from a third party (neurologist or a State based ALS organization) they must be willing to transfer care to the neurologist participating in the study.

Following completion of the 36-week randomized placebo controlled treatment period, interested participants must meet the following inclusion criteria to enroll in the open-label extension:

1. Participants must have completed the randomized placebo controlled Treatment Period without compliance issues
2. Able to understand and give written informed consent to participant in the open-label extension.
3. If referred from a third party (neurologist or a State based ALS organization), participant agrees to maintain transfer of care to a neurologist participating in the study.

Exclusion Criteria:

1. Patients will be excluded from the study if they meet any of the following criteria:
2. At Screening patients who utilize, or in the Investigator's judgment will be imminently dependent upon:

   1. Non-invasive ventilation > 22 hours per day, or
   2. Tracheostomy Note: If the patient requires non-invasive ventilation postrandomisation, they will be allowed to continue in the study.
3. Patients with Familial ALS (e.g., 2 or more family members with ALS or motor neuron disease)
4. Patients with a history of carpal tunnel syndrome, polyneuropathy, or in the investigators judgement diseases that could induce polyneuropathy and interfere with electromyography (EMG) recordings.
5. Patients with too severe atrophy of the Abductor Digiti Minimi (ADM), Abductor Pollicis Brevis (APB), Biceps Brachii (BB), or Tibialis Anterior (TA) muscles in the least clinically affected hand and leg, respectively, to allow for reliable EMG recordings.
6. Patient with a history of significant other major medical conditions based on the Investigator's judgment.
7. Based on the investigator's judgment, patients who may have difficulty complying with the protocol and/or any study procedures.
8. Patient with clinically significant abnormalities in haematology, blood chemistry, ECG, or physical examination not resolved by the Baseline visit which according to Investigator can interfere with study participation.
9. Patients with clinically significant hepatic or renal dysfunction or clinical laboratory findings that would limit the interpretability of change in liver or kidney function, or those with low platelet counts (< 150 x 109 per liter) or eosinophilia (absolute eosinophil count of ≥ 500 eosinophils per microliter) at Screening.
10. Patient participating in any other investigational drug trial or using investigational drug (within 12 weeks prior to screening and thereafter).
11. Females who are pregnant or nursing or who plan to get pregnant during the course of this clinical trial or within 6 months of the end of this trial.
12. Females of child-bearing potential, or men, who are unwilling or unable to use accepted methods of birth control.
13. Active inflammatory condition or autoimmune disorder.
14. Positive screen for drugs of abuse.
15. History of gold allergy.
16. Patient is considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator.

Following completion of the 36-week randomized placebo controlled treatment period, interested participants will be excluded from participating in the open-label extension phase if they meet any of the following criteria:

1. Lack of treatment compliance during the randomized placebo controlled Treatment Period.
2. Positive pregnancy test at the Week 36 visit, or, females who plan to get pregnant during the course of this extension or within 6 months of the end of this extension.
3. Based on the investigator's judgment, patients who may have difficulty complying with the protocol and/or any study procedures.
4. Patient with clinically significant abnormalities in hematology, blood chemistry, ECG, or physical examination identified during the W36 visit which according to Investigator may interfere with continued participation.
5. Patients with clinically significant hepatic or renal dysfunction or clinical laboratory.

   findings that would limit the interpretability of change in liver or kidney function, or those with low platelet counts (< 150 x 109 per liter) or eosinophilia (absolute eosinophil count of ≥ 500 eosinophils per microliter) at the Week 36 visit.
6. Patient is considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parvarthi Menon, PhD, MD, MBBS, Principal Investigator — Westmead Hospital; William Huynh, MD, Principal Investigator — University of Sydney, Brain and Mind Centre
Locations (2):
- Australia (2):
  - University of Sydney Brain and Mind Centre, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vucic S, Menon P, Huynh W, Mahoney C, Ho KS, Hartford A, Rynders A, Evan J, Evan J, Ligozio S, Glanzman R, Hotchkin MT, Kiernan MC. Efficacy and safety of CNM-Au8 in amyotrophic lateral sclerosis (RESCUE-ALS study): a phase 2, randomised, double-blind, placebo-controlled trial and open label extension. EClinicalMedicine. 2023 Jun 8;60:102036. doi: 10.1016/j.eclinm.2023.102036. eCollection 2023 Jun. PMID 37396808
- [Derived] Saha S, Tripathy S, Patra CR. Neuritogenic activity of metal nanoparticles. Nanomedicine (Lond). 2024 Feb;19(5):363-366. doi: 10.2217/nnm-2023-0297. Epub 2024 Jan 12. No abstract available. PMID 38214170
- [Derived] Vucic S, Kiernan MC, Menon P, Huynh W, Rynders A, Ho KS, Glanzman R, Hotchkin MT. Study protocol of RESCUE-ALS: A Phase 2, randomised, double-blind, placebo-controlled study in early symptomatic amyotrophic lateral sclerosis patients to assess bioenergetic catalysis with CNM-Au8 as a mechanism to slow disease progression. BMJ Open. 2021 Jan 11;11(1):e041479. doi: 10.1136/bmjopen-2020-041479. PMID 33431491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Phase 2, Randomised, Double-Blind, Placebo-Controlled Study in Early Symptomatic Amyotrophic Lateral Sclerosis Patients on Stable Background Therapy to Assess Bioenergetic Catalysis with CNM-Au8 to Slow Disease Progression in ALS. Recruitment started on December 19, 2019, with primary completion occurring on July 13, 2021. Participants enrolled at two institutional sites in Australia.
Pre-assignment Details: There was no washout or run-in period that occurred between ICF signing and IP initiation. Once the participant signed the ICF and was confirmed to be eligible for the study, they were randomized into the study and dosed with IP.
Groups:
- Placebo: The matched placebo used in this study consisted of water, sodium bicarbonate, and food coloring to match volume and color of the experimental treatment
  Placebo: Placebo is liquid with identical color and taste
Period: Overall Study
Arm/Group | Placebo | 30 mg CNM-Au8
Started | 22 | 23
Completed | 19 | 22
Not Completed | 3 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: The matched placebo to be used in this study will consist of water, sodium bicarbonate, and food coloring to match volume and color of the experimental treatment
  Placebo: Placebo is liquid with identical color and taste
- Total: Total of all reporting groups
Arm/Group | Placebo | 30 mg CNM-Au8 | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (10.89) | 57.0 (13.32) | 59.1 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 16 | 19 | 35
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Australia | 22 | 23 | 45
Height [Mean (Standard Deviation); unit: cm] | 167.2 (8.16) | 172.4 (11.81) | 169.9 (10.39)
Baseline Weight [Mean (Standard Deviation); unit: kg] | 69.2 (14.84) | 79.1 (18.09) | 74.3 (17.14)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (3.85) | 26.5 (4.86) | 25.5 (4.45)

OUTCOME MEASURES:

1. Primary Outcome: Electromyography Measures of Disease Progression.
Description: The Motor Unit Number Index (MUNIX) is a quantitative neurophysiological measure that provides an index of the number of lower motor neurons supplying a muscle. It reflects the loss of motor neurons in patients with ALS. Mean change in the average difference between active treatment and placebo from Baseline through Week 36 for the MUNIXscore(4), which is the sum of the respective MUNIX values for the Abductor Digiti Minimi (ADM), Abductor Pollicis Brevis (APB), Biceps Brachii (BB), and Tibialis Anterior (TA). The average baseline summed values will be indexed to 100%. Changes will be calculated as the percent change from the Baseline index of 100%.
Time Frame: 36 weeks
Population: Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 30 mg CNM-Au8
Number analyzed (Participants) | 22 | 23
percent change | -39.6 (7.1) | -31.8 (6.6)
Statistical Analysis 1: Comparison: Placebo vs 30 mg CNM-Au8; Test type: Superiority; p = 0.4304, MMRM; Mean Difference (Final Values) = 7.7, 95% CI 2-sided [-11.9 to 27.3]

2. Secondary Outcome: Percentage Mean Change in the Average Difference Between Active Treatment and Placebo From Baseline for Respiratory Function as Measured by Forced Vital Capacity (FVC).
Description: Mean change in FVC - Forced Vital Capacity.
Time Frame: 36 weeks
Population: Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 30 mg CNM-Au8
Number analyzed (Participants) | 22 | 23
percent change | -20.3 (5.8) | -16.7 (5.4)
Statistical Analysis 1: Comparison: Placebo vs 30 mg CNM-Au8; Test type: Superiority; p = 0.6519, MMRM; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-12.4 to 19.7]

3. Secondary Outcome: Mean Absolute Change of the Average Difference Between Active Treatment and Placebo From Baseline Through Week 36 for the MUNIXscore(4).
Description: The Motor Unit Number Index (MUNIX) is a quantitative neurophysiological measure that provides an index of the number of lower motor neurons supplying a muscle. It reflects the loss of motor neurons in patients with ALS. MUNIX will be reviewed via electromyography for the Abductor Pollicus Brevis (APB), Abductor Digiti Minimi (ADM), Biceps Brachii (BB), and Tibialis Anterior (TA). MUNIXscore(4) is the sum of the respective MUNIX values for the above mentioned muscle groups. A higher MUNIX value signifies greater muscle function. A greater decrease in the Mean absolute change signifies worsening muscle function.
Time Frame: 36 weeks
Population: Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: index score
Arm/Group | Placebo | 30 mg CNM-Au8
Number analyzed (Participants) | 22 | 23
index score | -141.3 (27) | -123.6 (25)
Statistical Analysis 1: Comparison: Placebo vs 30 mg CNM-Au8; Test type: Superiority; p = 0.6158, MMRM; Mean Difference (Final Values) = 18.8, 95% CI 2-sided [-56.4 to 94.0]

4. Other Pre Specified Outcome: Mean Change in the Average Difference Between Active Treatment and Placebo From Baseline Through Week 36 (Overall Difference at All Time Points) as Measured by MScanFit MUNE (Jacobsen et al., 2017) of the APB.
Description: The baseline average will be indexed to 100%, and changes at Week 12 and Week 36 will be calculated as the percent change from the Baseline index of 100%.
Time Frame: 36 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Mean Change in the Average Difference Between Active Treatment and Placebo From Baseline Through Week 36 for the MUSIXscore(4) (Neuwirth et al., 2015), Which is the Mean of the Respective MUSIX Values for the ADM, APB, BB, and TA.
Description: MUNIXscore(4) is the mean of the respective MUSIX values for the ADM, APB, BB, and TA. The average baseline mean values will be indexed to 100%. Changes will be calculated as the percent change from the Baseline index of 100%.
Time Frame: 36 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Mean Change in the Average Difference Between Active Treatment and Placebo From Baseline for the Neurophysiological Index (NPI) of the ADM.
Description: NPI is a method to quantify peripheral disease burden in ALS. NPI is defined as the ulnar nerve (ADM [CMAP peak amplitude] / ADM [distal motor latency]) x (ADM [f-wave %]).
Time Frame: 36 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Mean Change in the Average Difference Between Active Treatment and Placebo From Baseline for the Split Hand Index (SI).
Description: The SI is an early clinical feature that is used as a neurophysiological biomarker for evaluating ALS. Split Hand Index, defined as the first dorsal interosseous (FDI)Peak CMAP Amplitude * APBPeak CMAP Amplitude/ADMPeak CMAP Amplitude.
Time Frame: 36 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Mean Change in Average ALSFRS-R Score
Description: The ALS Functional Rating Scale-Revised (ALSFRS-R) is a validated rating instrument for monitoring the progression of disability in patients with ALS. Maximum score is 40, minimum is 0. A higher score signifies greater function.
Time Frame: 36 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 30 mg CNM-Au8
Number analyzed (Participants) | 22 | 23
score on a scale | -5.8 (0.9) | -4.8 (0.8)
Statistical Analysis 1: Comparison: Placebo vs 30 mg CNM-Au8; Test type: Superiority; p = 0.4249, MMRM; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-1.6 to 3.6]

9. Other Pre Specified Outcome: Mean Change Between Active Treatment and Placebo in the Proportion of Patients Experiencing a > 6-point Decline in the ALSFRS-R Between Active Treatment and Placebo.
Description: Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R)
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 30 mg CNM-Au8
Number analyzed (Participants) | 22 | 23
Participants
  Declined: Yes | 18 | 12
  Declined: No | 4 | 11
Statistical Analysis 1: Comparison: Placebo vs 30 mg CNM-Au8; Test type: Superiority; p = 0.0350, Chi-squared

10. Other Pre Specified Outcome: Mean Change in Slope of the Decline of the ALSFRS-R
Description: The ALS Functional Rating Scale-Revised (ALSFRS-R) is a validated rating instrument for monitoring the progression of disability in patients with ALS.
Time Frame: 36 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Mean Change Between Active Treatment and Placebo for the Combined Assessment of Function and Survival (CAFS), a Joint-rank Analysis of Function (ALSFRS-R) and Overall Survival
Description: the Combined Assessment of Function and Survival (CAFS). CAFS ranks patients' clinical outcomes based on survival time and change in the ALS Functional Rating Scale-Revised (ALSFRS-R) score. Each patient's outcome is compared to every other patient's outcome, assigned a score, and the summed scores are ranked. The mean rank score for each treatment group can then be calculated. A higher mean CAFS score indicates a better group outcome. There is no maximum or minimum due to ranking.
Time Frame: 36 weeks
Population: Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: Average change of rank
Arm/Group | Placebo | 30 mg CNM-Au8
Number analyzed (Participants) | 22 | 23
Average change of rank | -4.6 (5.2) | 4.4 (5.1)
Statistical Analysis 1: Comparison: Placebo vs 30 mg CNM-Au8; Test type: Superiority; p = 0.2237, ANCOVA; Mean Difference (Final Values) = 9.1, 95% CI 2-sided [-5.8 to 23.9]

12. Other Pre Specified Outcome: Time to ALS Clinical Worsening
Description: ALS Clinical Worsening is defined as the occurrence of death, tracheostomy, use of non-invasive ventilatory respiratory support, insertion of a gastrostomy tube, or a 6-point drop in the ALSFRS-R score. This outcome measures the number of participants that experienced ALS clinical worsening event within the 36 week time frame.
Time Frame: 36 weeks
Measure: Number; unit: participants
Arm/Group | Placebo | 30 mg CNM-Au8
Number analyzed (Participants) | 22 | 23
participants | 13 | 5
Statistical Analysis 1: Comparison: Placebo vs 30 mg CNM-Au8; Test type: Superiority; p = 0.0125, Log Rank; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.103 to 0.815]

13. Other Pre Specified Outcome: Mean Change in Rate of Disease Progression Defined as the Average Change in the Functional Survival (FS) Score ([Max ALSFRS-R Minus Current ALSFRS-R Score]/Symptom Duration in Months)
Description: Change in FS score = (Max ALSFRS-R minus current ALSFRS-R score) divided by symptom duration in months.
Time Frame: 36 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Mean Change in Average Difference Between Active Treatment and Placebo for the ALSSQOL-Short Form Questionnaire (ALSSQOL-SF)
Description: ALS Specific Quality of Life - Short Form (ALSSQOL-SF) Questionnaire will be completed at multiple times during the trial and the scores will be averaged. Maximum score is 10, minimum score is 0. A higher score signifies a higher quality of life.
Time Frame: 36 weeks
Measure: Least Squares Mean (Standard Error); unit: Average score on a scale
Groups:
- Placebo: The matched placebo to be used in this study consisted of water, sodium bicarbonate, and food coloring to match volume and color of the experimental treatment
  Placebo: Placebo is liquid with identical color and taste
Arm/Group | Placebo | 30 mg CNM-Au8
Number analyzed (Participants) | 22 | 23
Average score on a scale | -1.2 (0.3) | -0.3 (0.2)
Statistical Analysis 1: Comparison: Placebo vs 30 mg CNM-Au8; Test type: Superiority; p = 0.0177, MMRM; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [0.2 to 1.6]

15. Other Pre Specified Outcome: Mean Change in Average Difference Between Active Treatment and Placebo for the Clinician's Global Impression (CGI)
Description: The CGI scales (assessing both severity [CGI-S] and improvement [CGI-I]) provides a brief assessment of the clinician's view of the patient's global functioning and severity of current disease state and can be utilized to assess for changes in disease progression over the course of a clinical trial.
Time Frame: 36 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Mean Change in Average Difference Between Active Treatment and Placebo for the Patient's Global Impression (PGI)
Description: The PGI scales (assessing both severity [PGI-S] and improvement [PGI-I]) provides a brief assessment of the patient's view global functioning and severity of current disease state and can be utilized to assess for changes in disease progression over the course of a clinical trial.
Time Frame: 36 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Difference in the Proportion of Patients Utilizing Health Economic Outcome Measures
Time Frame: 36 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of the signing of the Informed Consent to 28 days after the last day of study drug administration, up to 46 weeks.
Arm/Group | Placebo | 30 mg CNM-Au8
All-Cause Mortality (participants affected / at risk) | 2/22 | 1/23
Serious Adverse Events (participants affected / at risk) | 5/22 | 5/23
Other Adverse Events (participants affected / at risk) | 17/22 | 17/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | 30 mg CNM-Au8 (N=23)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemorrhoids (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Motor neurone disease (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | 30 mg CNM-Au8 (N=23)
Fall (Injury, poisoning and procedural complications) | 3 | 2
Laceration (Injury, poisoning and procedural complications) | 3 | 0
Chest Injury (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Back Injury (Injury, poisoning and procedural complications) | 0 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Gingival discolouration (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Sweat gland infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Motor neurone disease (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastrostomy (Surgical and medical procedures) | 1 | 0
Myringotomy (Surgical and medical procedures) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT04098406/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT04098406/SAP_001.pdf